CLINICAL TRIAL: NCT05262335
Title: Anlotinib Plus Chemotherapy as First-line Therapy for Gastrointestinal Tumor Patients With Unresectable Liver Metastasis: A Multi-cohort, Multi-center Clinical Trial (ALTER-G-001)
Brief Title: Anlotinib Plus Chemotherapy as First-line Therapy for Gastrointestinal Tumor Patients With Unresectable Liver Metastasis (ALTER-G-001)
Acronym: ALTER-G-001
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021223
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-02

CONDITIONS: Gastrointestinal Tumors
MeSH Terms: conditions — Digestive System Neoplasms | interventions — anlotinib; Oxaliplatin; Capecitabine; Cisplatin; Paclitaxel; Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: Experimental group 1 (Experimental): Initial treatment: Anlotinib + Oxaliplatin + Capecitabine. Maintenance treatment (after 6 cycles): Anlotinib + Capecitabine
  Interventions: Drug: Anlotinib + Oxaliplatin + Capecitabine
- Experimental: Experimental group 2 (Experimental): Initial treatment: Anlotinib + Cisplatin + Paclitaxel/ Docetaxel. Maintenance treatment (after 6 cycles): Anlotinib + Capecitabine
  Interventions: Drug: Anlotinib + Cisplatin + Paclitaxel/ Docetaxel
- Experimental: Experimental group 3 (Experimental): Initial treatment: Anlotinib + Standard first-line chemotherapy Maintenance treatment (after 6 cycles): Anlotinib + Capecitabine
  Interventions: Drug: Anlotinib + Standard first-line chemotherapy

INTERVENTIONS:
Drug: Anlotinib + Oxaliplatin + Capecitabine — 1. Before 6 cycles, Anlotinib 12mg, po.qd, d1-14; Capecitabine 850 mg/m2, po. bid, d1-14; Oxaliplatin 130 mg/m2, iv (D1). The above schemes are repeated every three weeks.
  2. After 6 cycles, the regimen is changed to Anlotinib (12mg, po.qd, d1-14)+ Capecitabine (500 mg, po. bid, d1-21). The regimen is repeated every 3 weeks until the disease progresses or unacceptable toxicity.
  Arms: Experimental: Experimental group 1
Drug: Anlotinib + Cisplatin + Paclitaxel/ Docetaxel — 1. Anlotinib 12mg, po.qd, d1-14; Cisplatin 60-75mg/m2, iv, d1/d1-d3; Paclitaxel 135mg/m2, iv (D1). or Docetaxel 75mg/m2, iv (D1). The above schemes are repeated every three weeks.
  2. After 6 cycles, the regimen is changed to Anlotinib (12mg, po.qd, d1-14)+ Capecitabine (500 mg, po. bid, d1-21). The regimen is repeated every 3 weeks until the disease progresses or unacceptable toxicity.
  Arms: Experimental: Experimental group 2
Drug: Anlotinib + Standard first-line chemotherapy — 1. Anlotinib 12mg, po.qd, d1-14; Standard first-line chemotherapy determined by the researchers. The above schemes are repeated every three weeks.
  2. After 6 cycles, the regimen is changed to Anlotinib (12mg, po.qd, d1-14)+ Capecitabine (500 mg, po. bid, d1-21). The regimen is repeated every 3 weeks until the disease progresses or unacceptable toxicity.
  Arms: Experimental: Experimental group 3

SUMMARY:
This is an open, multi-cohort, multi-center, exploratory and phase II clinical trial. To evaluate the efficacy and safety Anlotinib combined with chemotherapy as first-line and maintenance therapy for Gastrointestinal Tumors with Unresectable Liver Metastases.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed Ⅳ phase of colorectal cancer with liver metastases (TanyNanyM1), and the liver metastases are unresectable; Or Histologically or cytologically confirmed Ⅳb phase of esophageal squamous cell carcinoma with liver metastases (TanyNanyM1) (excluding mixed type adenosquamous carcinoma), and the liver metastases are unresectable; Or Histologically or cytologically confirmed other gastrointestinal tumors with liver metastases (excluding gastrointestinal stromal tumors, neuroendocrine tumors and other malignant tumors of non-glandular epithelial origin), and the liver metastases are unresectable;
* No previous systemic treatment, including chemotherapy, targeted and immunotherapy;
* The target lesion must contain liver metastases. According to RECIST version 1.1, liver metastases have at least one measurable focus;
* Age from 18-75 years old;
* ECOG performance status of 0-1;
* Life expectancy of at least 3 months;
* The main organs are functioning normally (normal main organs function as defined below: Hemoglobin (Hb) ≥ 90 g/L, Neutrophils (ANC) ≥ 1.5×109/L, Platelet count (PLT) ≥ 90×109/L, Total bilirubin (TBIL) ≤ 1.5 × normal upper limit (ULN), Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 5 ×ULN, Creatinine Clearance rate (CCr) ≥60ml/min)
* Women of childbearing potential should agree to use and utilize an adequate method of contraception (such as intrauterine device，contraceptive and condom) throughout treatment and for at least 3 months after study is stopped；the result of serum or urine pregnancy test should be negative before enrollment；Man participants should agree to use and utilize an adequate method of contraception throughout treatment and for at least 2 months after study is stopped.
* Subjects volunteered to join the study, signed informed consent, good compliance, with follow-up.

Exclusion Criteria:

Patients with active bleeding within 2 months of primary and/or metastatic lesions;

* Patients with previous arterial/venous thrombosis events within 6 months, such as cerebrovascular accidents (including temporary ischemic attack), deep venous thrombosis or pulmonary embolism;
* Patients who are receiving thrombolytic or anticoagulant therapies such as warfarin, heparin, or their analogists; allowed to take low-dose heparin (6000 to 12,000 U/d for adults) or low-dose aspirin (≤100 mg/d) for prophylactic purposes with an INR≤1.5×ULN;
* Gastrointestinal diseases with a bleeding tendency (such as active gastrointestinal ulcer) or be likely to cause gastrointestinal bleeding, perforation, or obstruction, or patients with fistula;
* Have undergone major surgery (craniotomy, thoracotomy or open surgery) within 4 weeks prior to the first dose study;
* HER2-positive gastric adenocarcinoma;
* A history of immunodeficiency, including a positive HIV test or other acquired, congenital immunodeficiency disease, or a history of organ transplantation;
* A variety of factors affecting oral medications (such as inability to swallow, chronic diarrhea, and intestinal obstruction);
* Symptomatic central nervous system metastasis and/or cancerous meningitis are known to exist;
* Patients with any severe and / or uncontrolled disease, including: Patients with hypertension that cannot be well controlled by single antihypertensive therapy (SBP ≥150 mmHg, Diastolic BP ≥100mmHg); Or taking two or more antihypertensive drugs to control blood pressure; Acute myocardial infarction, malignant arrhythmias (including QT interval > 450ms in men and > 470ms in women) and ≥2 grade congestive heart failure (NYHA grade); Active or uncontrolled severe infection (NCI-CTC AE grade ≥2 infection); Liver diseases such as cirrhosis, decompensated liver disease, active hepatitis, or chronic hepatitis (HBV-DNA > 1000 IU/mL) require antiviral therapy; Diabetic patients with poor blood glucose control (fasting blood glucose (FBG) > 10 mmol/L); Routine urine indicated urine protein ≥ ++, and confirmed 24-hour urine protein quantitative > 1.0 g;
* Clinically significant ascites, including any ascites that can be found on a physical examination, ascites that has been treated or currently in need of treatment, and only those with a small amount of ascites but no symptoms can be selected;
* A moderate amount of fluid in both sides of the chest, or a large amount of fluid in one side of the chest, or has caused respiratory dysfunction Patient to be drained;
* Uncontrolled metabolic disorders or other non-malignant organs or secondary reactions to systemic diseases or cancers that may lead to higher medical risk and/or uncertainty in survival evaluation;
* Known to have active tuberculosis;
* Suffering from interstitial lung disease requiring steroid therapy;
* Significantly malnourished patients;
* Those who have a history of psychotropic substance abuse and are unable to quit or have a mental disorder;
* Known to be allergic to the test drug;
* Participated in clinical trials of other anti-tumor therapies within 4 weeks;
* Pregnant or lactating women.;
* History of other primary malignancies, but the following: 1) complete remission of malignant tumors for at least 2 years prior to enrollment and no additional treatment during the study; 2) non-melanoma skin cancer or malignant freckle-like sputum with adequate treatment and no evidence of disease recurrence; 3) adequately treated and In situ carcinoma without evidence of disease recurrence;
* According to the investigator's judgment, there are serious concomitant diseases that endanger the safety of the patient or affect the patient's completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 24 months
  Objective response rate is defined as the percentage of subjects whose best response was complete response (CR) or partial response (PR) according to the RECIST v1.1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 24 months
  Progression-free survival is defined as the time from enrollment to the date of first document disease progression or death from any cause.
Disease Control Rate (DCR) | up to 24 months
  Disease control rate is defined as the percentage of subjects whose best response was CR, PR or stable disease (SD) according to the RECIST v1.1.
Duration of Response (DoR) | up to 24 months
  Duration of Response is defined as the percentage of subjects whose best response was CR, PR or stable disease (SD) according to the RECIST v1.1 or death due to any cause, whichever occurs first.
Safety: Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Until 30 day safety follow-up visit
  Adverse events assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (version 5.0).
Overall Survival (OS) | Up to 24 months
  Overall Survival (OS) is defined as the time from enrollment to death from any cause.
Radical Resection Rate of Liver Metastases | Up to 6 cycles
  Radical Resection Rate of Liver Metastases is defined as the percentage of subjects whose liver metastases from unresectable to resectable.

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Jiannan University, Wuxi, Jiangsu
  - Wuxi Branch of Rujin Hospital, Wuxi, Jiangsu
  - Jiading Cental Hospital Shanghai University of Medicine & Health Sciences, Shanghai
  - Ruijin Hospital, Shanghai
  - Tongji Hospital of Tongji University, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu JW, Zhou CF, Han ZX, Zhang H, Yan J, Chen J, Wang CB, Qin ZQ, Mao Y, Tang XY, Zhu LJ, Wei XW, Cui DH, Yang XL, Shi M, Zhao LQ, Jiang JL, Zhu WY, Wang HM, Wang C, Zhu LJ, Zhang J. Anlotinib plus chemotherapy as a first-line treatment for gastrointestinal cancer patients with unresectable liver metastases: a multicohort, multicenter, exploratory trial. Signal Transduct Target Ther. 2024 Dec 9;9(1):344. doi: 10.1038/s41392-024-02051-4. PMID 39648217
- [Derived] Li H, Feng H, Zhang T, Wu J, Shen X, Xu S, Xu L, Wang S, Zhang Y, Jia W, Ji X, Cheng X, Zhao R. CircHAS2 activates CCNE2 to promote cell proliferation and sensitizes the response of colorectal cancer to anlotinib. Mol Cancer. 2024 Mar 21;23(1):59. doi: 10.1186/s12943-024-01971-7. PMID 38515149